CLINICAL TRIAL: NCT04286607
Title: A Phase 3, Multicenter, Open-Label Extension Study of the Long-Term Safety of ARQ-151 Cream 0.3% in Subjects With Chronic Plaque Psoriasis
Brief Title: Open-Label Extension Trial of PDE4 Inhibition With Roflumilast for the Management of Plaque Psoriasis
Acronym: DERMIS-OLE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Arcutis Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARQ-151-306
Record Dates: First submitted 2020-02-25; First posted 2020-02-27 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Chronic Plaque Psoriasis
MeSH Terms: interventions — Roflumilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ARQ-151 Cream 0.3% (Experimental)
  Interventions: Drug: Topical roflumilast

INTERVENTIONS:
Drug: Topical roflumilast — Active treatment
  Other Names: ARQ-151 Cream 0.3%

SUMMARY:
This study will assess the safety and efficacy of ARQ-151 cream applied once a day for 24 weeks by subjects with chronic plaque psoriasis

DETAILED DESCRIPTION:
This is an open-label study in which ARQ-151 cream is applied once daily x 24 weeks to subjects with psoriasis

ELIGIBILITY:
Inclusion Criteria:

* Participants legally competent to sign and give informed consent or informed consent of legal guardian, and, if age appropriate, assent by the subject, as required by local laws
* Males and females ages 2 years and older (inclusive)
* Subjects with chronic plaque psoriasis who meet eligibility criteria and:

  1. Successfully completed a prior ARQ-151 cream study in psoriasis (Cohort 1) or
  2. Are naïve to treatment with ARQ-151 cream (Cohort 2)
* Females of childbearing potential (FOCBP) must have a negative pregnancy test at all study visits. In addition, sexually active FOCBP must agree to use at least one form of highly effective contraception throughout the trial.

Exclusion Criteria:

* Subjects who experienced an ARQ-151 treatment-related AE or a serious AE (SAE) that precluded further treatment with ARQ-151 cream in a prior ARQ-151 cream study.
* Planned excessive exposure of treated area(s) to either natural or artificial sunlight, tanning bed or other LED.
* Females who are pregnant, wishing to become pregnant during the study, or are breast-feeding.
* Subjects with any serious medical condition or laboratory abnormality that would prevent study participation or place the subject at significant risk, as determined by the Investigator.
* Subjects with a history of chronic alcohol or drug abuse within 6 months of initiation of investigational product.
* Subjects who are unable to communicate, read or understand the local language, or who display another condition, which in the Investigator's opinion, makes them unsuitable for clinical study participation.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 333 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-01-22 (Actual)

PRIMARY OUTCOMES:
Occurrence of treatment emergent AEs (TEAEs) | 24 weeks
  The occurrence of TEAEs and the occurrence of (Serious Adverse Events) SAEs

SECONDARY OUTCOMES:
Achievement of an Investigator Global Assessment (IGA) of 'clear' or 'almost clear' over time. | 24 weeks
In subjects who achieve a 'clear' IGA time to re-starting investigational product (duration of response). | 24 weeks
Achievement of a 50% reduction in (Psoriasis Area Severity Index) PASI over time | 24 weeks
Achievement of a 75% reduction in PASI over time | 24 weeks
Achievement of a 90% reduction in PASI over time | 24 weeks
Achievement of a 100% reduction in PASI over time | 24 weeks
Change in Worst Itch Numeric Rating Scale) WI-NRS score over time | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David Berk, MD, Study Director — Arcutis Biotherapeutics, Inc.
Locations (85):
- United States (68):
  - Arcutis Biotherapeutics Clinical Site 203, Scottsdale, Arizona
  - Arcutis Biotherapeutics Clinical Site 239, Beverly Hills, California
  - Arcutis Biotherapeutics Clinical Site 127, Encinitas, California
  - Arcutis Biotherapeutics Clinical Site 225, Encino, California
  - Arcutis Biotherapeutics Clinical Site 509, Fountain Valley, California
  - Arcutis Biotherapeutics Clinical Site 112, Fremont, California
  - Arcutis Biotherapeutics Clinical Site 120, Irvine, California
  - Arcutis Biotherapeutics Clinical Site 508, Los Angeles, California
  - Arcutis Biotherapeutics Clinical Site 511, Rancho Santa Margarita, California
  - Arcutis Biotherapeutics Clinical Site 123, San Diego, California
  - Arcutis Biotherapeutics Clinical Site 220, San Diego, California
  - Arcutis Biotherapeutics Clinical Site 136, San Francisco, California
  - Arcutis Biotherapeutics Clinical Site 208, Santa Monica, California
  - Arcutis Biotherapeutics Clinical Site 215, Santa Monica, California
  - Arcutis Biotherapeutics Clinical Site 223, Boynton Beach, Florida
  - Arcutis Biotherapeutics Clinical Site 237, DeLand, Florida
  - Arcutis Biotherapeutics Clinical Site 118, Delray Beach, Florida
  - Arcutis Biotherapeutics Clinical Site 202, Hialeah, Florida
  - Arcutis Biotherapeutics Clinical Site 228, Largo, Florida
  - Arcutis Biotherapeutics Clinical Site 131, Miami, Florida
  - Arcutis Biotherapeutics Clinical Site 201, North Miami Beach, Florida
  - Arcutis Biotherapeutics Clinical Site 137, Ocala, Florida
  - Arcutis Biotherapeutics Clinical Site 105, Sanford, Florida
  - Arcutis Biotherapeutics Clinical Site 209, Sweetwater, Florida
  - Arcutis Clinical Site 602, Boise, Idaho
  - Arcutis Biotherapeutics Clinical Site 114, Plainfield, Illinois
  - Arcutis Biotherapeutics Clinical Site 102, Rolling Meadows, Illinois
  - Arcutis Biotherapeutics Clinical Site 214, Indianapolis, Indiana
  - Arcutis Biotherapeutics Clinical Site 217, Louisville, Kentucky
  - Arcutis Biotherapeutics Clinical Site 111, Baton Rouge, Louisiana
  - Arcutis Biotherapeutics Clinical Site 211, Lake Charles, Louisiana
  - Arcutis Biotherapeutics Clinical Site 213, Metairie, Louisiana
  - Arcutis Biotherapeutics Clinical Site 224, New Orleans, Louisiana
  - Arcutis Biotherapeutics Clinical Site 125, Rockville, Maryland
  - Arcutis Biotherapeutics Clinical Site 138, Rockville, Maryland
  - Arcutis Biotherapeutics Clinical Site 101, Brighton, Massachusetts
  - Arcutis Biotherapeutics Clinical Site 116, Clinton Township, Michigan
  - Arcutis Biotherapeutics Clinical Site 212, Detroit, Michigan
  - Arcutis Biotherapeutics Clinical Site 216, Fridley, Minnesota
  - Arcutis Biotherapeutics Clinical Site 227, Saint Joseph, Missouri
  - Arcutis Biotherapeutics Clinical Site 219, Las Vegas, Nevada
  - Arcutis Biotherapeutics Clinical Site 231, Las Vegas, Nevada
  - Arcutis Biotherapeutics Clinical Site 139, Reno, Nevada
  - Arcutis Biotherapeutics Clinical Site 240, Reno, Nevada
  - Arcutis Biotherapeutics Clinical Site 236, Portsmouth, New Hampshire
  - Arcutis Biotherapeutics Clinical Site 129, East Windsor, New Jersey
  - Arcutis Biotherapeutics Clinical Site 121, New York, New York
  - Arcutis Biotherapeutics Clinical Site 130, Rochester, New York
  - Arcutis Biotherapeutics Clinical Site 108, Stony Brook, New York
  - Arcutis Biotherapeutics Clinical Site 115, High Point, North Carolina
  - Arcutis Biotherapeutics Clinical Site 124, Fairborn, Ohio
  - Arcutis Biotherapeutics Clinical Site 222, Oklahoma City, Oklahoma
  - Arcutis Biotherapeutics Clinical Site 134, Oklahoma City, Oklahoma
  - Arcutis Biotherapeutics Clinical Site 229, Broomall, Pennsylvania
  - Arcutis Biotherapeutics Clinical Site 128, Duncansville, Pennsylvania
  - Arcutis Biotherapeutics Clinical Site 113, Exton, Pennsylvania
  - Arcutis Biotherapeutics Clinical Site 135, Pittsburgh, Pennsylvania
  - Arcutis Biotherapeutics Clinical Site 233, Knoxville, Tennessee
  - Arcutis Biotherapeutics Clinical Site 221, Murfreesboro, Tennessee
  - Arcutis Biotherapeutics Clinical Site 206, Arlington, Texas
  - Arcutis Biotherapeutics Clinical Site 104, College Station, Texas
  - Arcutis Biotherapeutics Clinical Site 119, Dallas, Texas
  - Arcutis Biotherapeutics Clinical Site 519, Frisco, Texas
  - Arcutis Biotherapeutics Clinical Site 238, Houston, Texas
  - Arcutis Biotherapeutics Clinical Site 110, San Antonio, Texas
  - Arcutis Biotherapeutics Clinical Site 117, San Antonio, Texas
  - Arcutis Biotherapeutics Clinical Site 210, West Jordan, Utah
  - Arcutis Biotherapeutics Clinical Site 230, Richmond, Virginia
- Canada (16):
  - Arcutis Biotherapeutics Clinical Site 132, Calgary, Alberta
  - Arcutis Biotherapeutics Clinical Site 207, Surrey, British Columbia
  - Arcutis Biotherapeutics Clinical Site 226, Surrey, British Columbia
  - Arcutis Biotherapeutics Clinical Site 232, Winnepeg, Manitoba
  - Arcutis Biotherapeutics Clinical Site 234, Fredericton, New Brunswick
  - Arcutis Biotherapeutics Clinical Site 205, Ajax, Ontario
  - Arcutis Biotherapeutics Clinical Site 218, Barrie, Ontario
  - Arcutis Biotherapeutics Clinical Site 103, London, Ontario
  - Arcutis Biotherapeutics Clinical Site 133, Mississauga, Ontario
  - Arcutis Biotherapeutics Clinical Site 140, Ottawa, Ontario
  - Arcutis Biotherapeutics Clinical Site 109, Peterborough, Ontario
  - Arcutis Biotherapeutics Clinical Site 235, Toronto, Ontario
  - Arcutis Biotherapeutics Clinical Site 106, Waterloo, Ontario
  - Arcutis Biotherapeutics Clinical Site 204, Windsor, Ontario
  - Arcutis Biotherapeutics Clinical Site 107, Montreal, Quebec
  - Arcutis Biotherapeutics Clinical Site 126, Québec, Quebec
- Arcutis Clinical Site 601, Santo Domingo, Dominican Republic